CLINICAL TRIAL: NCT03513016
Title: A Phase 1, Double-Blind, Randomized, Placebo Controlled, Single Ascending Dose Study to Assess the Safety and Tolerability of UBX0101 in Moderate to Severe, Painful Osteoarthritis of the Knee
Brief Title: A Safety and Tolerability Study of UBX0101 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Unity Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: UBX0101-OAR-101
Record Dates: First submitted 2018-04-27; First posted 2018-05-01 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Painful Osteoarthritis; Osteoarthritis, Knee; Senescence
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: UBX0101 (Experimental): Part A: UBX0101, single intra-articular injection, ascending dose
  Interventions: Drug: UBX0101
- Part A: Placebo (Placebo Comparator): Part A: Placebo, single intra-articular injection, ascending dose
  Interventions: Other: Placebo
- Part B: UBX0101 (Experimental): Part B: UBX0101, single intra-articular injection, fixed dose
  Interventions: Drug: UBX0101
- Part B: Placebo (Placebo Comparator): Part B: Placebo, single intra-articular injection, fixed dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: UBX0101 — Investigational drug intra-articular injection
  Arms: Part A: UBX0101; Part B: UBX0101
Other: Placebo — Diluent intra-articular injection
  Arms: Part A: Placebo; Part B: Placebo

SUMMARY:
A study to evaluate safety, tolerability, and pharmacokinetics of a single intra-articular injection of UBX0101 in patients diagnosed with painful osteoarthritis of the knee.

DETAILED DESCRIPTION:
This study is a phase 1, randomized, double-blind, placebo-controlled single ascending dose study that will evaluate safety, tolerability, and pharmacokinetics of UBX0101 in patients diagnosed with painful femoro-tibial osteoarthritis. The study consists of 2 parts: Part A is a single ascending dose study, whereas Part B is a single-dose study at a dose that has been determined to be safe and tolerable in Part A of the study.

In Part A, subjects will be randomly allocated to receive UBX0101 or placebo in 3:1 randomization by dose level (cohort), whereas in Part B subjects will be randomly allocated to receive UBX0101 or placebo in a 2:1 randomization.

The primary objective is to establish the safety and tolerability of UBX0101 given as a single intra-articular injection into the femoro-tibial joint of patients with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have the capacity to give informed consent and who are willing to comply with all study related procedures and assessments. Patients who do not have the legal capacity or medical competency to give written informed consent are not eligible for this study; consent via legally authorized representative will not be accepted
* Patients must be ≥ 40 and ≤ 85 years of age
* Patients using non-steroidal anti-inflammatory agent must be on a consistent regimen, dose, and medication for at least 8 weeks prior to enrollment
* Part A only: Ambulatory persons with osteoarthritis (OA) of the knee and baseline pain with a mean of ≥ 4 and ≤ 9 points on the 24-hour mean pain score (on the 11-point Numeric Rating Scale) for at least five of the seven days during the screening period.
* Part B only: Ambulatory persons with painful osteoarthritis (OA) of the knee for at least six months.
* Part B only: Patients with OA must have Kellgren-Lawrence scores 1 through 4 in the target knee
* Part B only: Patients must have a baseline pain ≥6 on the WOMAC Index pain subscale as derived from the KOOS.

Exclusion Criteria:

* Any condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation or prevent the Patient from fully participating in all aspects of the study
* Patients with clinically significant co-existing conditions of the cardiovascular, renal, gastrointestinal, respiratory, nervous, metabolic, or hematologic/ immune systems
* Patients with a history of diabetes mellitus according to the American Diabetes Association criteria or patients previously diagnosed by a qualified physician as having diabetes (American Diabetes Association Standards of Medical Care in Diabetes 2016)
* Patients with a history of cardiac rhythm disturbances, abnormal ECG intervals, or use of medications known to impact ECG intervals
* Patients who have undergone diagnostic arthroscopy of the Target Knee in the previous six months
* Patients who have undergone arthroscopic surgery in the last two years prior to the screening visit (including microfracture and menisectomy) on the Target Knee.
* Patients anticipated to have arthroscopic surgery on either knee at any time during the study period
* History of previous total or partial knee arthroplasty in either knee
* Part A only: Patients with an effusion at the screening visit which, in the opinion of the investigator following examination and discussions with the Patient, requires drainage for symptom relief
* Patients who have received intra-articular treatment with steroids or hyaluronic acid derivatives within the last 16 weeks prior to screening
* Patients who use, or have used in the 8 weeks prior to screening, opioid analgesics (with exception of mild opioid analgesics)
* Patients who have had regenerative joint procedures on any joint including, but not limited to, platelet-rich plasma injections, mesenchymal stem cell transplantation, autologous chondrocyte transplantation, or mosaicplasty
* Current or history of other joint diseases such as joint dysplasia, crystal-induced arthropathy (such as gout, or calcium pyrophosphate deposition disease evidenced by clinical and/or radiographic means), aseptic osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, or neuropathic arthropathy of any cause
* Any active known or suspected systemic autoimmune disease (except for vitiligo, residual auto-immune hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment for two years, conditions not expected to recur in the absence of an external trigger) or any history of a systemic inflammatory arthritis such as psoriatic, rheumatoid, ankylosing spondylitis or reactive arthritis
* Patients diagnosed presently and symptomatic with fibromyalgia based on American College of Radiology (ACR) Criteria
* Patients with a BMI ≥ 40 kg/m2, or whose size exceed the limits of the of the MRI equipment (coil and gantry)

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single intra articular injection of UBX0101 evaluated by the incidence of serious and non-serious adverse events | 12 weeks

SECONDARY OUTCOMES:
Part A: Plasma concentration of UBX0101 over 24 hrs following a single intra-articular injection | 24 hrs
Part A: The change from baseline to Week 12 of the weekly mean of the average daily pain intensity score as obtained using the 11-point numerical rating scale [0-10] where 0 represents no pain and 10 represents worst pain imaginable | Baseline to Week 12
Part A: The change from baseline to Week 12 for the Western Ontario and McMaster Universities (WOMAC) index total score and the pain and function subscales using the 5-point Likert scale | Baseline to Week 12
Part B: The change from baseline to Week 4 of selected senescence-associated secretory phenotype factors in plasma samples and in synovial fluid aspirates in patients receiving a single intra-articular injection of UBX0101 versus those receiving placebo. | Baseline to Week 4
Part B: The change from baseline to Week 4 for the Western Ontario and McMaster Universities (WOMAC) index pain subscale using as derived from Knee injury and Osteoarthritis Outcome Score (KOOS). | Baseline to Week 4
Part B: Plasma concentration of UBX0101 following a single intra-articular injection | 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Dananberg, MD, Study Chair — UNITY Biotechnology
Locations (7):
- United States (7):
  - TriWest Research Associates, El Cajon, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Well Pharma Medical Research, Miami, Florida
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - Clinical Research Consortium, Las Vegas, Nevada
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas